CLINICAL TRIAL: NCT04140279
Title: Effect of Latanoprostene Bunod Ophthalmic Solution 0.024% on Episcleral Venous Pressure and Outflow Facility in Ocular Hypertensive Subjects
Brief Title: A Study to Evaluate the Effect of Latanoprostene Bunod Ophthalmic Solution 0.024% on Episcleral Venous Pressure and Outflow Facility in Participants With Ocular Hypertension
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It never started
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 899
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Ocular Hypertension
Keywords: Eye Diseases
MeSH Terms: conditions — Ocular Hypertension; Eye Diseases | interventions — BOL 303259-X

STUDY DESIGN:
Intervention Model Description: All participants will receive both the investigational and placebo treatments, with 1 eye receiving LBN 0.024% and the contralateral eye receiving placebo.
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Latanoprostene Bunod (Experimental): Participants will receive LBN ophthalmic solution 0.024% in the applicable eye identified during randomization. The first dose will be instilled in the morning (AM) at approximately 11 AM on Day 1 and the remaining 6 doses will be instilled once per day in the evening at approximately 8 PM.
  Interventions: Drug: Latanoprostene Bunod
- Placebo (Placebo Comparator): Participants will receive Renu MultiPlus Lubricating and Rewetting Drops (placebo) in the applicable eye identified during randomization. The first dose will be instilled in the morning (AM) at approximately 11 AM on Day 1 and the remaining 6 doses will be instilled once per day in the evening at approximately 8 PM.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Latanoprostene Bunod — Ophthalmic solution
  Other Names: Vyzulta®
  Arms: Latanoprostene Bunod
Drug: Placebo — Ophthalmic solution, no active ingredient.
  Other Names: Bausch + Lomb ReNu MultiPlus® Lubricating and Rewetting Drops
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of latanoprostene bunod (LBN) ophthalmic solution 0.024% (a single dose and 7 days of once daily [QD] dosing) on 2 aspects of aqueous humor (AqH) dynamics (episcleral venous pressure [EVP] and outflow facility) in participants with ocular hypertension (OHT).

DETAILED DESCRIPTION:
All participants will receive both the investigational (LBN ophthalmic solution 0.024%) and placebo treatments, with 1 eye receiving LBN 0.024% and the contralateral eye receiving placebo. Each participant will be randomized as to which eye (right or left) will receive LBN 0.024% versus placebo.

All participants will undergo a minimum 14-day to maximum 42-day washout period prior to the start of study drug administration.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Participants must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB) approved informed consent form (ICF) and are able and willing to comply with all treatment and follow-up/study procedures.
* Females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must agree to use an acceptable method of contraception throughout their participation in the study.

Ocular Inclusion Criteria

* Participants must have a diagnosis of OHT in both eyes (intraocular pressure [IOP] ≥22 mmHg prior to starting treatment with IOP-lowering medication) without evidence of glaucomatous optic neuropathy or visual field loss and must also have been receiving IOP-lowering medication for ≥3 months prior to Screening (Visit 1).
* Participants must undergo a washout of any existing ocular hypotensive medications in order to determine eligibility. Washout period will vary with the class of medication used (2-6 weeks).
* Participants must meet the following IOP requirements at Visit 3 (Eligibility Visit at End of Washout):

  1. Intraocular pressure ≥22 mmHg and ≤32 mmHg in both eyes.
  2. An increase in IOP of 20% over the Screening (Visit 1) IOP.
  3. The difference in IOP between eyes ≤4 mmHg.
* Participants must have a best corrected visual acuity (BCV A) in each eye of 20/50 (logarithm of the minimum angle of resolution [logMAR] +0.4) or better.

Exclusion Criteria:

General Exclusion Criteria

* Participation in any drug or device clinical investigation within 30 days prior to Visit 1 (Screening) or anticipation of participating in any other drug or device clinical investigation within the duration of this study.
* Participants with a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the participant or confound the results of the study.
* Female participants who are pregnant or breastfeeding.

Drug Therapies

* Participants with an anticipated need to initiate or modify medication (systemic or topical) that is known to affect IOP (for example, steroids, α-adrenergic agonists, β-adrenergic antagonists, calcium channel blockers, angiotensin-converting enzyme [ACE] inhibitors, and angiotensin II receptor blockers).
* Participants with known hypersensitivity or contraindications to latanoprostene bunod or any of the ingredients in the study drugs.

Ocular Exclusion Criteria:

Diseases

* Participants who are unable to discontinue contact lens use during and for 15 minutes following instillation of study drug and for 24 hours before check-in and during each study visit.
* Participants with a central corneal thickness less than 480 μm or greater than 600 micrometer (μm) in either eye.
* Participants with any condition that prevents reliable applanation tonometry (for example, significant corneal surface abnormalities) in either eye.
* Participants who are monocular.
* Participants with ocular conditions, which, in the opinion of the Investigator, will impact the study measurements, such as:

  1. Active optic disc hemorrhage in either eye.
  2. Current or a history of central/branch retinal vein or artery occlusion in either eye.
  3. Current or a history of macular edema in either eye.
  4. Very narrow angles (3 quadrants with less than Grade 2 according to Shaffer's anterior chamber angle grading system) and participants with angle closure, congenital, and secondary glaucoma, and with history of angle closure in either eye.
  5. Diagnosis of a clinically significant or progressive retinal disease (for example, diabetic retinopathy, exudative or severe non-exudative macular degeneration) in either eye.
* Participants with any intraocular infection or inflammation in either eye within 3 months prior to Visit 1 (Screening).
* Myopia greater than -4.00 diopter (D), or hyperopia greater than +2.000

Surgery

* Participants with a history of ocular laser surgery in either eye within the 3 months (90 days) prior to Visit 1 (Screening).
* Participants with a history of laser trabeculoplasty, cyclophotocoagulation or glaucoma surgical procedures at any time prior to Visit 1 (Screening).
* Participants with a history of incisional ocular surgery other than routine uncomplicated cataract surgery or severe trauma in either eye within the 3 months (90 days) prior to Visit 1 (Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-13 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Episcleral Venous Pressure (EVP) at Intervals on Days 1 and 8 | Baseline, 1, 3, and 5 hours post-instillation at Day 1 and 12, 16, and 20 hours post-instillation at Day 8
  EVP will be measured non-invasively by using a custom-designed slit-lamp mounted venomanometer. This device utilizes the pressure chamber technique, in which a clear flexible balloon is placed against the surface of the eye, and the pressure is increased until an episcleral vein is noted to blanche. Each EVP measurement will be determined from the mean of up to 3 readings. EVP (millimeters of mercury [mmHg]) will be assessed at 1, 3, and 5 hours post instillation for changes from baseline following a single dose of drug on the first day of treatment and at approximately 12, 16 and 20 hours post-instillation after 7 days of QD in the evening treatment.
Change From Baseline in Diurnal (Daytime) EVP at Days 1 and 8 | Baseline, Day 1, Day 8
  EVP will be measured non-invasively by using a custom-designed slit-lamp mounted venomanometer. This device utilizes the pressure chamber technique, in which a clear flexible balloon is placed against the surface of the eye, and the pressure is increased until an episcleral vein is noted to blanche. Each EVP measurement will be determined from the mean of up to 3 readings. Diurnal EVP will be computed for Days 1 and 8 separately as the mean of the posttreatment values observed on the day for each eye. Change from the mean of 2 sets of baseline measurements will be computed for each post-treatment time (including diurnal means) as the post-treatment value minus the baseline value for each eye. The difference between treatments (LBN minus placebo) in change from baseline will be computed for each participant.
Change From Baseline in Trabecular Outflow Facility at Intervals on Days 1 and 8 | Baseline, 1, 3, and 5 hours post-instillation at Day 1 and 12, 16, and 20 hours post-instillation at Day 8
  Outflow facility will be measured non-invasively by using constant weight tonography. Four-minute tracings with a 5.5-gram or 7.5-gram weight or two-minute tracings with a 10-gram weight will be used, and tonographic outflow facility will be calculated from the pressure decay curves and standard tables. Outflow facility (mmHg) will be assessed at 1, 3, and 5 hours post instillation for changes from baseline following a single dose of drug on the first day of treatment and at approximately 12, 16 and 20 hours post-instillation after 7 days of QD in the evening treatment.
Change From Baseline in Diurnal (Daytime) Trabecular Outflow Facility at Days 1 and 8 | Baseline, Day 1, Day 8
  Outflow facility will be measured non-invasively by using constant weight tonography. Four-minute tracings with a 5.5-gram or 7.5-gram weight or 2-minute tracings with a 10-gram weight will be used, and tonographic outflow facility will be calculated from the pressure decay curves and standard tables. Diurnal trabecular outflow facility will be computed for Days 1 and 8 separately as the mean of the posttreatment values observed on the day for each eye. Change from the mean of 2 sets of baseline measurements will be computed for each post-treatment time (including diurnal means) as the post-treatment value minus the baseline value for each eye. The difference between treatments (LBN minus placebo) in change from baseline will be computed for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch Site 001, Rochester, Minnesota, United States